CLINICAL TRIAL: NCT03250117
Title: An Open-Label, Relative Bioavailability Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Ropinirole Implants in Patients With Parkinson's Disease Switched From Oral Immediate-Release Ropinirole While on L-Dopa
Brief Title: Relative Bioavailability Study of Ropinirole Implants in Parkinson's Patients on L-Dopa Switched From Oral Ropinirole
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated for reasons not related to efficacy or safety
Sponsor: Titan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ROP-001
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Dyskinesia; ropinirole; implant; ProNeura; movement disorders; dopamine agonist; extended-release; Parkinsonian disorders; brain diseases; central nervous system diseases; Neurodegenerative Diseases; Antiparkinson agents; Anti-dyskinesia agents; dopamine agents; neurotransmitter agents; REQUIP; subdermal
MeSH Terms: conditions — Parkinson Disease; Dyskinesias; Movement Disorders; Parkinsonian Disorders; Brain Diseases; Central Nervous System Diseases; Neurodegenerative Diseases | interventions — ropinirole

STUDY DESIGN:
Intervention Model Description: Subjects receive oral immediate release (IR) ropinirole for 7-10 days, and then are switched to ropinirole implant(s) for 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Requip; One Ropinirole Implant
  Interventions: Drug: Ropinirole oral product; Drug: Ropinirole Implant
- Cohort 2 (Experimental): Requip; Two Ropinirole Implants
  Interventions: Drug: Ropinirole oral product; Drug: Ropinirole Implant
- Cohort 3 (Experimental): Requip; Three Ropinirole Implants
  Interventions: Drug: Ropinirole oral product; Drug: Ropinirole Implant
- Cohort 4 (Experimental): Requip; Four Ropinirole Implants
  Interventions: Drug: Ropinirole oral product; Drug: Ropinirole Implant

INTERVENTIONS:
Drug: Ropinirole oral product — oral immediate-release ropinirole
  Other Names: Requip
Drug: Ropinirole Implant — ropinirole hydrochloride/ethylene vinyl acetate

SUMMARY:
Subjects stable on L-Dopa and oral ropinirole will have their ropinirole replaced with the Ropinirole Implant(s). The Ropinirole Implant was designed using the ProNeura™ implant technology where the implant is inserted under the skin. This study will measure how much ropinirole is released in the blood during 12 weeks of ropinirole implant treatment, and evaluate the side effects of this new formulation.

ELIGIBILITY:
Key Inclusion Criteria:

* Voluntarily provided informed consent
* Meet diagnostic criteria for idiopathic Parkinson's Disease
* On L-Dopa and oral ropinirole
* If female of child-bearing potential, willing to practice contraception from time of informed consent to Follow-Up Visit

Key Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant
* Active epilepsy within the past year
* Severe dementia or cognitive impairment
* Donated or lost > 400 mL of blood within 1 month prior to Screening
* History of alcohol or substance use disorder within the prior 12 months
* Recent episodes of moderate to severe dizziness or syncope
* Definite or suspected hypersensitivity to ropinirole or ethylene vinyl acetate
* Used any other investigational drug within 60 days or 5 half-lives prior to Screening, or plan to take any such drug any time during the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kate Beebe DeVarney, Study Director — Titan Pharmaceuticals
Locations (3):
- United States (3):
  - Orlando, Florida, Orlando, Florida
  - Farmington Hills, Michigan, Farmington Hills, Michigan
  - Kirkland, Washington, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 6 screened patients, 3 did not meet eligibility criteria for cohort assignment.
Period: Requip IR [7-10 Days]
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 3 | 0 (Study terminated before cohort opened to enrollment) | 0 (Study terminated before cohort opened to enrollment) | 0 (Study terminated before cohort opened to enrollment)
Completed | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Ropinirole Implant 12 Weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 3 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — At request of Sponsor, regulatory agencies, or the IRB | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 52.7 [47 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
MDS-UPDRS Total Score [Mean (Full Range); unit: units on a scale] — Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Scale [MDS-UPDRS] is a questionnaire and examination rating motor and non-motor experiences, and motor complications. Score is summed to range from 0 to 272. Higher score indicates more severe symptoms/outcome.
  units on a scale | 60.7 [23 to 97]
Awake Time "On" [Mean (Full Range); unit: hours] — Diaries were completed for 2 consecutive days prior to the visit, used to record motor state in half-hour intervals over a 24-hour period (during waking hours). "On" refers to when medication is providing benefit with regard to mobility, slowness and stiffness, regardless of dyskinesia. Daily totals for waking hours were normalized to a 16-hour waking day and averaged across the 2 days.
  hours | 11.54 [9.9 to 14.3]
Awake Time "Off" [Mean (Full Range); unit: hours] — Diaries were completed for 2 consecutive days prior to the visit, used to record motor state in half-hour intervals over a 24-hour period (during waking hours). "Off" refers to when medication has worn off and is no longer providing benefit with regard to mobility, slowness and stiffness. Daily totals for waking hours were normalized to a 16-hour waking day and averaged across the 2 days.
  hours | 5.02 [3.4 to 6.1]

OUTCOME MEASURES:

1. Primary Outcome: AUC0-24 Hours of Ropinirole
Description: Area under the plasma drug concentration-time curve of ropinirole
Time Frame: 0-24 hours
Population: Subjects who received at least 1 ropinirole implant and for whom at least 1 PK parameter of interest can be calculated were to be included in this analysis. Analysis not performed due to insufficient representative samples from each cohort.
Arm/Group | Cohort 1
Number analyzed (Participants) | 0

2. Primary Outcome: Total Number of Adverse Events Across Participants
Description: Safety and tolerability of ropinirole implant(s) presented as the total number of adverse events experienced by the analysis population.
Time Frame: 0-12 weeks
Population: Subjects who received a least 1 ropinirole implant
Measure: Number; unit: Events
Arm/Group | Cohort 1
Number analyzed (Participants) | 3
Events | 4

3. Secondary Outcome: AUC0-24 Hours of N-despropyl Ropinirole
Description: Area under the plasma drug concentration-time curve of N-despropyl ropinirole
Time Frame: 0-24 hours
Population: as for outcome 1
Arm/Group | Cohort 1
Number analyzed (Participants) | 0

4. Secondary Outcome: AUC0-24 Hours of 7-hydroxy Ropinirole
Description: Area under the plasma drug concentration-time curve of 7-hydroxy ropinirole
Time Frame: 0-24 hours
Population: as for outcome 1
Arm/Group | Cohort 1
Number analyzed (Participants) | 0

5. Secondary Outcome: Mean Change From Baseline in MDS-UPDRS Total Score
Description: Efficacy of ropinirole implants presented as the mean change from baseline in MDS-UPDRS total score. Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Scale [MDS-UPDRS] is a questionnaire and examination rating motor and non-motor experiences, and motor complications. Score is summed to range from 0 to 272. Higher score indicates more severe symptoms/outcome.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: Subjects who receive at least 1 ropinirole implant and complete at least 1 post-baseline efficacy assessment. Three subjects were in the analysis population at Week 4. Two subjects were in the analysis population at Weeks 8 and 12.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort 1
Number analyzed (Participants) | 3
units on a scale
  Week 4 | 4.0 (3.28)
  Week 8 | 10.6 (13.42)
  Week 12 | 7.3 (4.04)

6. Secondary Outcome: Mean Change From Baseline of Awake Time "On"
Description: Efficacy of ropinirole implants presented as mean change from baseline of awake time "on". Diaries were completed for 2 consecutive days prior to the visit, used to record motor state in half-hour intervals over a 24-hour period (during waking hours). "On" refers to when medication is providing benefit with regard to mobility, slowness and stiffness, regardless of dyskinesia. Daily totals for waking hours were normalized to a 16-hour waking day and averaged across the 2 days.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, 8, 10, 12
Population: Subjects who receive at least 1 ropinirole implant and complete at least 1 post-baseline efficacy assessment. Three subjects were in the analysis population for Weeks 1-6. Two subjects were in the analysis population for Weeks 8-12.
Measure: Mean (Standard Error); unit: hours
Arm/Group | Cohort 1
Number analyzed (Participants) | 3
hours
  Week 1 | 0.80 (1.078)
  Week 2 | 1.11 (0.457)
  Week 3 | 1.70 (0.908)
  Week 4 | 0.77 (0.608)
  Week 6 | 0.66 (1.175)
  Week 8 | 0.11 (1.344)
  Week 10 | 0.93 (0.756)
  Week 12 | 0.58 (1.101)

7. Secondary Outcome: Mean Change From Baseline of Awake Time "Off"
Description: Efficacy of ropinirole implants presented as mean change from baseline of awake time "Off". Diaries were completed for 2 consecutive days prior to the visit, used to record motor state in half-hour intervals over a 24-hour period (during waking hours). "Off" refers to when medication has worn off and is no longer providing benefit with regard to mobility, slowness and stiffness. Daily totals for waking hours were normalized to a 16-hour waking day and averaged across the 2 days
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, 8, 10, 12
Population: as for outcome 6
Measure: Mean (Standard Error); unit: hours
Arm/Group | Cohort 1
Number analyzed (Participants) | 3
hours
  Week 1 | -1.36 (0.974)
  Week 2 | -1.67 (0.921)
  Week 3 | -2.26 (1.062)
  Week 4 | -1.33 (1.094)
  Week 6 | -1.22 (1.506)
  Week 8 | -0.83 (2.068)
  Week 10 | -1.77 (1.598)
  Week 12 | -1.43 (1.943)

ADVERSE EVENTS:
Time Frame: From signing of the ICF until 30 days following study drug treatment discontinuation, up to 22 weeks.
Description: Subjects assessed for AEs at every visit, routine collection of safety labs, and spontaneous self-reporting.
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3)
Implant site reaction (General disorders) | 1 (1)
Freezing phenomenon (Nervous system disorders) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a first-in-human study of ropinirole implants. The trial was terminated early at the request of the Sponsor, not for reasons of safety or efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has rights to first publication of results unless waived by Sponsor. PIs may publish following Sponsor first publication or 18 months after conclusion, abandonment or termination of study. Sponsor to review proposed publications prior to public release and can embargo results for up to 60 days from the time submitted to the Sponsor for review and may remove any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT03250117/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT03250117/SAP_001.pdf